CLINICAL TRIAL: NCT03563001
Title: Differences of Small Airways Function Between Chronic Obstructive Pulmonary Disease(COPD) and Asthma-copd Overlap(ACO)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-HXNK-002
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome; Small Airway Disease; Quality of Life
Keywords: chronic obstructive pulmonary disease; asthma-chronic obstructive pulmonary disease overlap; small airway; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome | interventions — Budesonide; Formoterol Fumarate; BID protein, human; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Patients with diagnosis of simple chronic obstructive pulmonary disease(COPD) and asthma-chronic obstructive pulmonary disease overlap(ACO) are recruited.Small airways function of subjects in both group(chronic obstructive pulmonary disease and asthma-chronic obstructive pulmonary disease overlap) is assessed at baseline.And then budesonide(160ug) and formoterol(4.5ug) bid will be given to the subjects for 3 months.The subjects will have a follow-up visit with the same examinations after 3 months' treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Obstructive Pulmonary Disease Group (Experimental): Patients with diagnosis of chronic obstructive pulmonary disease according to Global Initiative for Chronic Obstructive Disease(GOLD 2018) are recruited.Small airways function of is assessed at baseline.And then budesonide(160ug) and formoterol(4.5ug) bid will be given to the subjects for 3 months.The subjects will have a follow-up visit with the same examinations after 3 months' treatment.
  Interventions: Drug: Budesonide(160ug) and Formoterol(4.5ug) bid
- Asthma-Chronic Obstructive Pulmonary Disease Overlap Group (Experimental): Patients with diagnosis of asthma-chronic obstructive pulmonary disease overlap according to Global Initiative for Chronic Obstructive Disease(GOLD 2018),Global Initiative for Asthma(GINA 2018) and Spanish COPD Guidelines(GesEPOC 2017) are recruited.Small airways function of is assessed at baseline.And then budesonide(160ug) and formoterol(4.5ug) bid will be given to the subjects for 3 months.The subjects will have a follow-up visit with the same examinations after 3 months' treatment.
  Interventions: Drug: Budesonide(160ug) and Formoterol(4.5ug) bid

INTERVENTIONS:
Drug: Budesonide(160ug) and Formoterol(4.5ug) bid — For both groups of subjects,small airways function of is assessed at baseline.And then budesonide(160ug) and formoterol(4.5ug) bid will be given to the subjects for 3 months.The subjects will have a follow-up visit with the same examinations after 3 months' treatment.
  Other Names: SYMBICORT TURBUHALER

SUMMARY:
The purpose of this study is to research the differences of small airways function between subjects with diagnosis of chronic obstructive pulmonary disease(COPD) and asthma-COPD overlap(ACO).The assessment of quality of life is also carried out through questionnaires.

DETAILED DESCRIPTION:
This is a randomized,open-label study to research the differences of small airways function between simple chronic obstructive pulmonary disease(COPD) and asthma-COPD overlap(ACO).Assessment of small airways is conducted at baseline,including forced expired volume in one second(FEV1),forced vital capacity(FVC),peak expiratory flow(PEF),maximum expiratory flow rate at 75% of vital capacity(MEF75),maximum expiratory flow rate at 50% of vital capacity(MEF50),maximum expiratory flow rate at 25% of vital capacity(MEF25),impulse oscillometry,diffusion function,residual volume(RV) and total lung capacity(TLC).Budesonide(160ug) and formoterol(4.5ug) bid will be given to both groups(chronic obstructive pulmonary disease and asthma-COPD overlap) for 3 months.Quality of life is assessed through questionnaires including modified Medical Research Council dyspnoea scale(mMRC),St George's Respiratory Questionnaire(SGRQ) and chronic obstructive pulmonary disease assessment test(CAT).All of the patients will have a follow-up visit after 3 months' treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 to 80 years-old.
* A diagnosis of chronic obstructive pulmonary disease according to the Global Initiative for Chronic Obstructive Disease(GOLD 2018) guidelines are recruited to the chronic obstructive pulmonary disease group.A diagnosis of asthma-chronic obstructive pulmonary disease overlap according to Global Initiative for Chronic Obstructive Disease(GOLD 2018),Global Initiative for Asthma(GINA 2018) and Spanish COPD Guidelines(GesEPOC 2017) are recruited to the asthma-chronic obstructive pulmonary disease overlap group.
* Willing and able to provide written informed consent.
* Willing and able to attend all study visits and adhere to all study assessments and procedures.

Exclusion Criteria:

* Severe comorbidities including unstable cardiac or pulmonary disease or any other medical conditions including unstable ischemic heart disease,unstable cardiac arrhythmia or heart failure,life threatening arrhythmias,etc.
* Recent history of chronic obstructive pulmonary disease exacerbation requiring hospitalization or need for increased treatments for chronic obstructive pulmonary disease within 6 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Differences of maximum expiratory flow rate at 75% of vital capacity(MEF75) between chronic obstructive pulmonary disease and asthma-chronic obstructive pulmonary disease overlap | 3 months
  Maximum expiratory flow rate at 75% of vital capacity(MEF75) is measured according to internationally accepted standards in both groups by Jaeger MasterScreen Pulmonary Function Test System.

SECONDARY OUTCOMES:
Differences of maximum expiratory flow rate at 50% of vital capacity(MEF50) between two groups | 3 months
  Maximum expiratory flow rate at 50% of vital capacity(MEF50) is measured according to internationally accepted standards in both groups by Jaeger MasterScreen Pulmonary Function Test System.
Differences of maximum expiratory flow rate at 25% of vital capacity(MEF25) between two groups | 3 months
  Maximum expiratory flow rate at 25% of vital capacity(MEF25) is measured according to internationally accepted standards in both groups by Jaeger MasterScreen Pulmonary Function Test System.
Differences of impulse oscillometry parameters between two groups | 3 months
  Impulse oscillometry parameters are measured according to internationally accepted standards in both groups by Jaeger MasterScreen Pulmonary Function Test System.
Differences of diffusion function between two groups | 3 months
  Diffusion function is measured according to internationally accepted standards in both groups by Jaeger MasterScreen Pulmonary Function Test System.
Differences of residual volume(RV) between two groups | 3 months
  Residual volume(RV) is measured according to internationally accepted standards in both groups by Jaeger MasterScreen Pulmonary Function Test System.
Differences of total lung capacity(TLC) between two groups | 3 months
  Total lung capacity(TLC) is measured according to internationally accepted standards in both groups by Jaeger MasterScreen Pulmonary Function Test System.
Changes of maximum expiratory flow rate at 75% of vital capacity(MEF75) after 3 months' treatment compared with baseline in both groups | Change from baseline to 3 months
  At baseline,maximum expiratory flow rate at 75% of vital capacity(MEF75) is performed in each subject.After 3 months's treatment of budesonide and formoterol,the test will be performed again.
Changes of maximum expiratory flow rate at 50% of vital capacity(MEF50) after 3 months' treatment compared with baseline in both groups | Change from baseline to 3 months
  At baseline,maximum expiratory flow rate at 50% of vital capacity(MEF50) is performed in each subject.After 3 months's treatment of budesonide and formoterol,the test will be performed again.
Changes of maximum expiratory flow rate at 25% of vital capacity(MEF25) after 3 months' treatment compared with baseline in both groups | Change from baseline to 3 months
  At baseline,maximum expiratory flow rate at 25% of vital capacity(MEF25) is performed in each subject.After 3 months's treatment of budesonide and formoterol,the test will be performed again.
Changes of impulse oscillometry parameters(IOS) after 3 months' treatment compared with baseline in both groups | Change from baseline to 3 months
  At baseline,impulse oscillometry is performed in each subject.After 3 months's treatment of budesonide and formoterol,the test will be performed again.
Changes of diffusion function after 3 months' treatment compared with baseline in both groups | Change from baseline to 3 months
  At baseline,diffusion function is performed in each subject.After 3 months's treatment of budesonide and formoterol,the test will be performed again.
Changes of total lung capacity(TLC) after 3 months' treatment compared with baseline in both groups | Change from baseline to 3 months
  At baseline,total lung capacity(TLC) is performed in each subject.After 3 months's treatment of budesonide and formoterol,the test will be performed again.
Changes of residual volume(RV) after 3 months' treatment compared with baseline in both groups | Change from baseline to 3 months
  At baseline,residual volume(RV) is performed in each subject.After 3 months's treatment of budesonide and formoterol,the test will be performed again.
Change of St George's Respiratory Questionnaire(SGRQ) scores after 3 months' treatment compared with baseline | Change from baseline to 3 months
  The SGRQ questionnaire is developed to measure the quality of life in patients with chronic airway diseases.Scores range from 0 to 100,higher scores indicates worse respiratory condition.The St George's Respiratory Questionnaire is performed in both groups at baseline.After 3 months's treatment of budesonide and formoterol,the scores will be measured again.
Change of modified Medical Research Council dyspnoea scale(mMRC) scores after 3 months' treatment compared with baseline | Change from baseline to 3 months
  The mMRC scale is used to assess the degree of breathlessness.The scores range from 0 to 4,higher scores indicates more serious respiratory condition.The mMRC is performed in both groups at baseline.After 3 months's treatment of budesonide and formoterol,the scores will be measured again.
Change of chronic obstructive pulmonary disease assessment test(CAT) after 3 months' treatment compared with baseline | Change from baseline to 3 months
  The CAT test is used to assess the impact of COPD on patients' daily life.The scores range from 0 to 40,higher scores indicates worse respiratory condition.The CAT test is performed in both groups at baseline.After 3 months's treatment of budesonide and formoterol,the test will be performed again.

CONTACTS AND LOCATIONS:
Overall Officials: Huapeng Yu, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China